CLINICAL TRIAL: NCT03595553
Title: A Phase 3, Randomized, Double-blind, Active Controlled Study to Compare the Efficacy and Safety of Ridinilazole (200 mg, Bid) for 10 Days With Vancomycin (125 mg, Qid) for 10 Days in the Treatment of Clostridium Difficile Infection (CDI)
Brief Title: Comparison of Ridinilazole Versus Vancomycin Treatment for Clostridium Difficile Infection
Acronym: Ri-CoDIFy 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMT19969/C004; NCT03595566 (obsolete NCT alias)
Record Dates: First submitted 2018-06-11; First posted 2018-07-23 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides difficile; Clostridium difficile; C. difficile; C. diff
MeSH Terms: conditions — Clostridium Infections | interventions — ridinilazole; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In both arms patients receive the same number of doses per day. Placebo tablets are included to maintain same number and appearance of IP in both arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ridinilazole (Experimental): ridinilazole 200mg bid
  Interventions: Drug: Ridinilazole
- vancomycin (Active Comparator): vancomycin 125 mg qid
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Ridinilazole — ridinilazole (200 mg bid)
  Other Names: 2,2'-di(pyridin-4-yl)-1H,1'H-5,5'-bi(benzimidazole), 2,2'-bis(4-pyridyl)-3H,3'H-5,5'-bibenzimidazole, 2-pyridin-4-yl-6-(2-pyridin-4-yl-3H-benzimidaz
  Arms: ridinilazole
Drug: Vancomycin — vancomycin (125 mg qid)
  Arms: vancomycin

SUMMARY:
Summit is developing ridinilazole as a novel antimicrobial for Clostridioides difficile Infection (CDI), formerly known as Clostridium difficile Infection, with the goal of demonstrating an improved Sustained Clinical Response rate in subjects treated with ridinilazole as compared to subjects treated with vancomycin.

A phase 2 proof of concept study, with vancomycin as comparator, demonstrated these attributes with a comparable safety profile. A high fecal concentration of ridinilazole and little systemic exposure were noted.

The rationale for this phase 3 study is to confirm the improvement in sustained clinical response of CDI over vancomycin and to compare the safety and tolerability of ridinilazole to that of vancomycin.

Ridinilazole plasma concentration will be assessed in a subset of patients.

ELIGIBILITY:
Inclusion Criteria

Patients are eligible to be included in the study only if all the following criteria apply:

1. Patient must be at least 18 years of age, at the time of signing the informed consent.
2. Have signs and symptoms of CDI including diarrhea such that in the Investigator's opinion, CDI antimicrobial therapy is required. Diarrhea is defined as a change in bowel habits, with ≥3 unformed bowel movements (UBMs) (5, 6 or 7 on the Bristol Stool Chart) in the 24 h prior to randomization.
3. Have the presence of either toxin A and/or B of C. difficile in the stool determined by a positive free toxin test (using a Sponsor agreed test). The stool sample must be current (produced within 72 hours prior to randomization).
4. Male or Female

   Male patients:

   • A male patient must agree to use contraception as detailed in Section 10.4 of this protocol during the treatment period and for at least 30 days after the last dose of study treatment and refrain from donating sperm during this period.

   Female patients:

   • A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: i. Not a woman of childbearing potential (WOCBP) OR ii. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study treatment.
5. Has provided documented signed informed consent and any authorizations required by local law (e.g. Protected Health Information [PHI]). If unable to read, understand and sign the informed consent form a legally authorized representative (LAR) may provide consent on the patient's behalf if permitted by the Institutional Review Board (IRB)/Ethics Committee (EC).

Exclusion Criteria

Patients are excluded from the study if any of the following criteria apply:

1. Have had more than one prior episode of CDI in the previous 3 months or more than 3 episodes in the past 12 months prior to randomization.
2. Have a history of chronic diarrheal disease including inflammatory bowel disease (Crohn's disease or ulcerative colitis).
3. Have had a positive diagnostic test for other GI pathogens, considered to be clinically relevant, within 2 weeks of randomization.
4. Have had major gastrointestinal (GI) surgery (e.g. significant bowel resection) within 3 months of randomization (this does not include appendectomy). The presence of a colostomy or ileostomy or likely requirement of an ostomy during the study.
5. Have life threatening or fulminant CDI with evidence of hypotension, septic shock, peritoneal signs or absence of bowel sounds, or toxic megacolon.
6. History of bone marrow or hematopoietic stem cell transplant at any time or a known current history of a severely compromised/suppressed immune system that, in the opinion of the Investigator, would make the patient unsuitable for the study.
7. Have had more than the equivalent of 24 hours of dosing of antimicrobial treatment active against the current episode of CDI prior to randomization. (i.e. more than four doses of oral vancomycin, two doses of fidaxomicin or three doses of metronidazole).
8. Prior or current use of anti-toxin antibodies including bezlotoxumab within the past 6 months prior to randomization.
9. Are unable to discontinue products used affecting disease progression at randomization.
10. Has been involved in a clinical trial and received an investigational medicinal product for indications other than CDI within 1 month or five half-lives (whichever is longer) or within 3 months if the investigational medical product was for CDI.
11. Have received an investigational vaccine against C. difficile.
12. Patients that the Investigator feels are inappropriate for the study this would include those;

    1. with any other condition that, in the Investigator's judgment, would make the patient unsuitable for inclusion in the study.
    2. who, in the opinion of the Investigator, are not likely to complete the study for whatever reason, e.g. short life expectancy.
    3. with known hypersensitivity or intolerance to ridinilazole, vancomycin, and/or their excipients
    4. who are unwilling or unable to comply with protocol requirements, e.g. complete the full course of study treatment per schedule, attend study visits, report diarrhea/suspected recurrence, provide stool samples, ingest capsules/tablets or blood draws.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Styles, MD, Study Director — Summit Therapeutics
Locations (149):
- United States (49):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - GI Alliance - Arizona Digestive Health - Sun City, Sun City, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - Paradigm Clinical Research Centers, Inc, Redding, California
  - University Of California Davis, Sacramento, California
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Alliance Medical Research LLC, Lighthouse PT, Florida
  - Phoenix Medical Research LLC, Miami, Florida
  - San Marcus Research, Miami Lakes, Florida
  - Gasteroenterology Group of Naples, Naples, Florida
  - HeuerMD Research Inc, Orlando, Florida
  - Pines Care Research Center Inc., Pembroke Pines, Florida
  - Bardmoor Gastroenterology, Seminole, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida
  - Florida Medical Clinic P.A., Zephyrhills, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Grand Teton Research Group PLLC, Idaho Falls, Idaho
  - GI Alliance - Illinois Gastro Group - Glenview, Glenview, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UnityPoint Health Peoria/Proctor, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - St. Vincent Hospital, Worcester, Massachusetts
  - Harper Hospital Department of Pharmacy Services, Detroit, Michigan
  - Detroit Receiving Hospital Department of Pharmacy Services, Detroit, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Revival Research Institute, LLC., Southfield, Michigan
  - Mercury Street Medical Group PLLC, Butte, Montana
  - AB Clinical Trials, Las Vegas, Nevada
  - New York Presbyterian Hospital Weill Cornell, New York, New York
  - James J. Peters VAMC, The Bronx, New York
  - ECU Adult Specialty Care, Greenville, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Chattanooga Research and Medicine CHARM, Chattanooga, Tennessee
  - GI Alliance - Texas Digestive Disease Consultants - Arlington, Arlington, Texas
  - GI Alliance - Texas Digestive Disease Consultants - Cedar Park, Cedar Park, Texas
  - DM Clinical Research (Conroe Regional Hospital), Conroe, Texas
  - FMC Science, Lampasas, Texas
  - GI Alliance - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - GI Alliance - Texas Digestive Disease Consultants - Webster, Webster, Texas
  - Infectious Diseases Associates of Central VA, Lynchburg, Virginia
- Argentina (6):
  - Centro Médico Talar, El Talar, Buenos Aires
  - Instituto Medico Platense, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Ramos Mejía, Buenos Aires
  - Hospital Privado Centro Medico Cordoba, Córdoba
  - Instituto Medico ALAS, Salta
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Mater Misericordiae, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Center, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Brazil (8):
  - Unidade de Pesquisa - NCS - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Santa Casa De Misericordia De Belo Horizonte, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
- Bulgaria (5):
  - MHAT "Sv.Ivan Rilski-2003"OOD, Dupnitsa, Kyustendil
  - "MHAT - Blagoevgrad, EOOD Department of Gastroenterology", Blagoevgrad
  - DCC1-Sliven Ltd., Sliven
  - DCC Alexandrovska, Sofia
  - Medical center - Izgrev, Sofia
- Canada (7):
  - Foothills Medical Centre, South Tower, Calgary, Alberta
  - Moncton Hospital/Horizon Health Network, Moncton, New Brunswick
  - Lakeridge Health, Oshawa, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux de la Mauricie-et-du-Centre-du-Quebec, Trois-Rivières, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec- ULaval, Québec
  - Recherche Médicale St-Jérôme Inc, Québec
- Greece (8):
  - General Hospital of Athens ''Evangelismos', Athens
  - General Hospital of Athens ''Alexandra'', Athens
  - "Pathophysiology Department Athens University Medical School", Athens
  - " ATTIKON University Hospital", Athens
  - "'Hygeia'' Hospital 2nd Department of Medicine and Infectious Diseases", Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Patras, Pátrai
  - ''Tzaneio'' General Hospital of Piraeus, Piraeus
- Hungary (11):
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház, Infektológia-Hepatológia Osztály, Gyula, Bekes County
  - Pest Megyei Flór Ferenc Kórház, V. Belgyógyászat, Kistarcsa, Pest County
  - Dr. Kenessey Albert Kórház Rendelőintézet, Tüdőgyógyászati Aktív Osztály, Balassagyarmat
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház IV. Belgyógyászat - 2. Gasztroenterológia, Békéscsaba
  - "Dél-Pesti Centrumkórház-OHII Szent László Kórház Infektológiai Osztály ", Budapest
  - Országos Korányi Pulmonológiai Intézet, Központi Intenzív osztály, Budapest
  - CRU Hungary Kft BAZ Megyei Kórház és Egyetemi Oktatókórház, Szent Ferenc Tagkórház, Miskolc
  - "Pécsi Tudományegyetem I. sz. Belgyógyászat i Klinika, Infektológiai tanszék", Pécs
  - Pécsi Tudományegyetem Klinikai Központi Gyógyszertár, Pécs
  - Csongrad County Dr. Bugyi Istvan Hospital, Dept. Of Internal Medicine, Szentes
  - Javorszy Odon Hospital, Vác
- New Zealand (3):
  - Waitemata District Health Board WDHB North Shore Hospital, Takapuna, Auckland
  - Taranaki District Health Board TDHB - Taranaki Base Hospital, New Plymouth, Taranki
  - Waikato District Health Board Waikato Hospital, Hamilton, Waikato Region
- Poland (12):
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów, Podkarpackie Voivodeship
  - SP ZOZ w Bochni Szpital Powiatowy im. B. Marty Wieckiej, Bochnia
  - Szpital Bocheński SP ZOZ w Bochni, Bochnia
  - Klinika Chorób Zakaźnych i Hepatologii Wojewódzki Szpital Obserwacyjno-Zakaźny im. Tadeusza Browicza, Bydgoszcz
  - Szpital Specjalistyczny w Chorzowie, Chorzów
  - Szpital Zakonu Bonifratrów, Katowice
  - Specjalistyczne Gabinety Sp z o.o., Krakow
  - Korczowski Bartosz Gabinet, Rzeszów
  - ENDOSKOPIA Sp. z o.o., Sopot
  - Centralny Szpital Kliniczny MSWiA Klinika Chorób Wewnętrznych i Gastroenterologii, Warsaw
  - Klinika Chorób Wewnętrznych i Gastroenterologii z Pododdziałem Leczenia Nieswoistych Chorób Zapalnych Jelit Centralny Szpital Kliniczny MSWiA, Warsaw
  - Wojewódzki Szpital Specjalistyczny im. J. Gromkowskiego we Wrocławiu; I Oddział Chorób Zakaźnych, Wroclaw
- Romania (9):
  - SUUMC-Boli infectioase, Bucharest
  - Clinical Hospital of Infectious and Tropical Diseases "Dr. Victor Babes", Bucharest
  - S.C. Sana Monitoring Srl, Bucharest
  - Spitalul Clinic de Boli Infectioase si Tropicale, Bucharest
  - Spitalul Minicipal Caracal, Caracal
  - Spitalul Clinic de Boli Infectioase Constanta, Constanța
  - Spitalul Clinic de Boli Infectioase- Sfanta Parascheva, Iași
  - Spitalul Clinic de Boli Infectioase, Iași
  - Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
- Russia (2):
  - " State Budgetary Institution of Healthcare "City Clinical Hospital of n.a. V.M.Buyanova" ", Moscow
  - State budget healthcare institution of Novosibirsk region "City clinical hospital #2", Novosibirsk
- South Korea (15):
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Wonju Severance Christian Hospital, Ilsan-dong, Gangwondo
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Hanyang University Seoul Hospital, Ansan, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Anyang-si, Seoul
  - Kyungpook National University Hospital, Daegu, Seoul
  - Yeungnam University Medical Center, Daegu, Seoul
  - Samsung Medical Center, Irwon-dong, Seoul
  - Keimyung University Dongsan Hospital, Daegu, Yeongnam
  - Inje University Seoul Paik Hospital, Junggu
  - Kangbuk Samsung Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Soeul
  - Asan Medical Center, Soeul
- Spain (8):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía. Hospital Provincial, Córdoba
  - "Hospital Universtiario Donostia ", Donostia / San Sebastian
  - Hospital General Universitario Gregorio Marañon, Madrid
  - "Hospital Universitario Marqués de Valdecilla ", Santander
  - Hospital Universitario de Balme, Seville
  - Hospital Universitari Sant Joan de Reus, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okhuysen PC, Ramesh MS, Louie T, Kiknadze N, Torre-Cisneros J, de Oliveira CM, Van Steenkiste C, Stychneuskaya A, Garey KW, Garcia-Diaz J, Li J, Duperchy E, Chang BY, Sukbuntherng J, Montoya JG, Styles L, Clow F, James D, Dubberke ER, Wilcox M. A Randomized, Double-Blind, Phase 3 Safety and Efficacy Study of Ridinilazole Versus Vancomycin for Treatment of Clostridioides difficile Infection: Clinical Outcomes With Microbiome and Metabolome Correlates of Response. Clin Infect Dis. 2024 Jun 14;78(6):1462-1472. doi: 10.1093/cid/ciad792. PMID 38305378
- [Derived] Carlson TJ, Endres BT, Basseres E, Gonzales-Luna AJ, Garey KW. Ridinilazole for the treatment of Clostridioides difficile infection. Expert Opin Investig Drugs. 2019 Apr;28(4):303-310. doi: 10.1080/13543784.2019.1582640. Epub 2019 Feb 26. PMID 30767587

RESULTS

PARTICIPANT FLOW:
Groups:
- Ridinilazole: ridinilazole (200 mg bid), coated tablet, oral route of administration.
- Vancomycin: vancomycin (125 mg qid), hard capsule, oral route of administration.
Period: Overall Study
Arm/Group | Ridinilazole | Vancomycin
Started | 370 | 375
Completed | 312 | 327
Not Completed | 58 | 48
Not completed — Withdrawal by Subject | 20 | 8
Not completed — Physician Decision | 3 | 2
Not completed — Adverse Event | 2 | 5
Not completed — Death | 24 | 22
Not completed — Lost to Follow-up | 6 | 7
Not completed — Other as indicated in CSR | 3 | 3
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridinilazole | Vancomycin | Total
Number analyzed (Participants) | 370 | 375 | 745
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 209 | 213 | 422
  >=65 years | 161 | 162 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (17.89) | 59.6 (17.42) | 59.4 (17.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 227 | 436
  Male | 161 | 148 | 309
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 60 | 100
  Not Hispanic or Latino | 322 | 305 | 627
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 11 | 10 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 16 | 26
  White | 333 | 331 | 664
  More than one race | 8 | 8 | 16
  Unknown or Not Reported | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 81 | 87 | 168
  Canada | 12 | 17 | 29
  Europe | 229 | 220 | 449
  Mexico | 5 | 11 | 16
  Brazil | 3 | 10 | 13
  Chile | 2 | 3 | 5
  Argentina | 1 | 0 | 1
  Peru | 1 | 0 | 1
  Israel | 17 | 15 | 32
  South Korea | 10 | 9 | 19
  Australia | 6 | 2 | 8
  New Zealand | 3 | 1 | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.64 (5.729) | 26.36 (5.732) | 26.54 (5.748)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Clinical Response (SCR) Defined as Clinical Response and no Recurrence of CDI Through 30 Days Post End of Treatment (EOT).
Description: This primary outcome measures the number of participants with Sustained Clinical Response (SCR). SCR is defined as Clinical Response and no recurrence of CDI through 30 days post End of Treatment (EOT). At D40, D70 and D100 the Investigator or medically qualified designee will determine if the patient has a sustained clinical response or experienced RECURRENCE since the previous assessment. The Investigator will assess cure/failure and recurrence based on available information which includes, but is not limited to, improvement from baseline in the number of UBMs, signs & symptoms of CDI, and the requirement for CDI medication. The Investigator should assess cure/failure in a way that best reflects the Investigator's standard clinical practice.
Time Frame: Day 40
Measure: Count of Participants; unit: Participants
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 370 | 375
Participants
  SCR based on Clinical Cure | 238 | 225
  SCR based on Clinical Cure Failure | 132 | 150

2. Secondary Outcome: Clinical Response
Description: defined as
  * less than 3 unformed bowel movements (UBMs) for consecutive days and maintained through EOT without further CDI treatment at EOT + 2 days, or
  * the investigator's assessment that the subject no longer needs specific CDI antimicrobial treatment after completion of the course of study medication.
Time Frame: Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 370 | 375
Participants
  Clinical Response | 320 | 346
  Clinical Response Failure | 50 | 29

3. Secondary Outcome: Clinical Cure
Description: defined as the resolution of diarrhea (<3 UBMs in the 1-day period immediately prior to EOT, that is maintained for 2 days after EOT).
Time Frame: Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 370 | 375
Participants
  Clinical Cure | 275 | 292
  Clinical Cure Failure | 95 | 83

4. Secondary Outcome: Sustained Clinical Response Over 60 Days
Description: defined as Clinical Response and no recurrence of CDI through 60 days post EOT
Time Frame: Day 70
Measure: Count of Participants; unit: Participants
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 370 | 375
Participants
  Sustained Clinical Response 60 Days Post EOT | 262 | 258
  Sustained Clinical Response 60 Days Post EOT Failure | 108 | 117

5. Secondary Outcome: Sustained Clinical Response Over 90 Days
Description: defined as Clinical Response and no recurrence of CDI through 90 days post EOT
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 370 | 375
Participants
  Sustained Clinical Response 90 Days Post EOT | 259 | 249
  Sustained Clinical Response 90 Days Post EOT Failure | 111 | 126

6. Secondary Outcome: Relative Abundance of the 3 Main Bile Acid Groups (Conjugated Primary, Primary and Secondary Bile Acids) From Baseline to EOT.
Description: This secondary outcome measures the relative abundance of the 3 main Bile Acid Groups (Conjugated Primary, Primary and Secondary Bile Acids) from Baseline to EOT.
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: percentage of abundance
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 370 | 375
percentage of abundance
  Secondary Bile Acid Group at Baseline | 33.34 (35.68) | 30.25 (34.13)
  Secondary Bile Acid Group at EOT | 38.13 (39.63) | 7.87 (22.69)
  Primary Bile Acid Group at Baseline | 55.03 (34.06) | 57.44 (33.08)
  Primary Bile Acid Group at EOT | 55.99 (38.06) | 65.72 (33.90)
  Conjugated Primary Bile Acid Group at Baseline | 11.64 (21.93) | 12.31 (21.56)
  Conjugated Primary Bile Acid Group at EOT | 5.88 (15.50) | 26.42 (31.62)

7. Secondary Outcome: Percentage of Change of α-diversity (Shannon Index) of the Microbiota in Stool Samples From Baseline to EOT.
Description: This secondary outcome measures the percentage of change of α-diversity (Shannon Index) of the microbiota in stool samples from baseline to EOT. Shannon index is a weighted statistic measuring both species richness and evenness. The Shannon Index is calculated by taking the relative abundance of each species and sums the relative abundance times the natural log of the relative abundance for each species. The value is converted into a positive value by times minus one. A higher Shannon Index means higher diversity
Time Frame: Day 10
Measure: Mean (95% Confidence Interval); unit: percent change in Shannon Index
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 272 | 280
percent change in Shannon Index | 37.06 [6.01 to 68.11] | -7.32 [-16.61 to 1.97]

8. Secondary Outcome: Measure of β-diversity of the Gut Microbiota Between Baseline and EOT Stool Samples (Bray-Curtis Index/Dissimilarity).
Description: This secondary outcome measures the β-diversity of the gut microbiota in stool samples from baseline to EOT. Bray-Curtis index/dissimilarity measures how different two samples are in the microbiome composition. The Bray-Curtis dissimilarity is graded between 0 and 1, where 0 means the two samples have the same composition (that is they share all the species and every species has the same abundance), and 1 means the two samples do not share any species.
Time Frame: Day 10
Measure: Mean (95% Confidence Interval); unit: Bray-Curtis Index
Arm/Group | Ridinilazole | Vancomycin
Number analyzed (Participants) | 272 | 280
Bray-Curtis Index | 0.7 [0.68 to 0.72] | 0.81 [0.79 to 0.83]

ADVERSE EVENTS:
Time Frame: All Serious Adverse Events (SAEs) will be collected from the signing of the informed consent form (ICF) until the D100 End of Study visit. All AEs will be collected from the time and date of first dose of study treatment until the D40 follow-up visit.
Description: The number of participants (both arms: ridinilazole and vancomycin) in Participant Flow module is different than the Adverse Event Results. The Participant Flow module reflects mITT population, whereas Adverse Event Results population reflects Safety Population. mITT Population patients did not have positive free toxin/CCNA Test and/or >=3 UBM at Baseline. Safety Population only requires treated subjects.
Groups:
- RIDINILAZOLE 200 MG: RIDINILAZOLE 200mg bid, coated tablet, oral route of administration.
- VANCOMYCIN 125 MG: VANCOMYCIN 125mg qid, hard capsule, oral route of administration.
Arm/Group | RIDINILAZOLE 200 MG | VANCOMYCIN 125 MG
All-Cause Mortality (participants affected / at risk) | 26/374 | 24/377
Serious Adverse Events (participants affected / at risk) | 32/374 | 30/377
Other Adverse Events (participants affected / at risk) | 124/374 | 117/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIDINILAZOLE 200 MG (N=374) | VANCOMYCIN 125 MG (N=377)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HCoV-OC43 infection (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIDINILAZOLE 200 MG (N=374) | VANCOMYCIN 125 MG (N=377)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 7 (7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3)
Asthenia (General disorders) | 2 (3) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (2)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0)
Blood potassium increased (Investigations) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Cytomegalovirus test positive (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 21 (21) | 14 (15)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (4) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemodialysis complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 5 (6) | 9 (9)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Immobile (Social circumstances) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (11) | 3 (3)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0)
Presbyopia (Eye disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (9) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Torulopsis infection (Infections and infestations) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT03595553/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT03595553/SAP_001.pdf